CLINICAL TRIAL: NCT07291882
Title: Serum Hyperbilirubinemia as an Early Predictive Factor for Complicated Appendicitis: Single Center Experience
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Asaad AbdelRahman AbdelAziz Ahmad, Director and lecturer of general surgery, Minia University
Other Study IDs: Serum Hyperbilirubinemia
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Appendicitis, Surgery
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simple appendicitis ( group A): Patients where no perforation, gangrene, or other complications were found during surgery.
  Interventions: Procedure: Appendectomy
- Complicated appendicitis (group B): • Complicated appendicitis group (B): Patients who presented with perforation or gangrene, confirmed via operative findings and histopathological examination.
  Total bilirubin levels was measured preoperatively as part of the routine laboratory workup.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Total bilirubin levels was measured preoperatively as part of the routine laboratory workup. Appendectomy done for all patients followed by histopathological evaluation of the excised appendix.

SUMMARY:
Serum total bilirubin provides a practical guide to early assessment of suspected appendicitis, supporting faster and more proportionate decisions-earlier escalation when overall risk is high and safe observation when it is low. Because testing is rapid, inexpensive, and universally available, integration into local diagnostic pathways is feasible.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with right iliac fossa pain diagnosed clinically as acute appendicitis and had undergone appendectomy

Exclusion Criteria:

* patients with past history of jaundice
* patients with history of hyperbilirubinemia hemolytic disease
* positive hepatitis viruses
* cholelithiasis
* acquired or congenital biliary disease
* cancer of the hepatobiliary system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting with acute appendicitis at the Minia university hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
measurement of serum total bilirubin in each case of appendicitis to clarify the relationship between serum hyperbilirubinemia and complicated appendicitis | between September 2024 and August 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No